CLINICAL TRIAL: NCT04446533
Title: Assessment of a Filming Formulation of Hydrogen Peroxide and Hyaluronic Acid (BMG0703) in the Treatment of Periodontitis, Compared to Placebo and 0.2% Chlorhexidine. A Randomised Controlled Clinical Trial.
Brief Title: Effect of a Hydrogen-Peroxide and Hyaluronic-Acid Mouthwash (BMG0703) in the Treatment of Periodontitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Milan (Other)
Collaborators: BMG Pharma (Industry)
Responsible Party: Principal Investigator, Chiara Occhipinti, Professor, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Orto_BMG0703_PRD_June_2020
Record Dates: First submitted 2020-06-16; First posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Periodontitis; Bleeding Gum; Pocket, Periodontal
Keywords: Periodontitis; Bleeding Gum; Periodontal Pocket
MeSH Terms: conditions — Periodontitis; Gingival Hemorrhage; Periodontal Pocket | interventions — Hydrogen Peroxide; Chlorhexidine

STUDY DESIGN:
Intervention Model Description: Following a professional oral hygiene session, subjects will be divided into three groups: BMG0703, active comparator a nd placebo.
  First application of products will be applied clinically, and subsequently, one bottle of the product (test, comparative or placebo) will be given to the patient to use it 3 times a day, after meals and after normal oral hygiene procedures, for at least one week.
  The subjects will then be re-evaluated after 3 days and after a week. During these check-ups, new samples will be collected at the level of the initial sampling sites and will be reassessed on the basis of the selected clinical indices (in particular plaque, bleeding and probing depth).
Who Masked: Participant, Investigator
Masking Description: The products will be packaged in such a way that they are not recognizable either by the operator or by the patient. Each package will be assigned a number that in turn will refer to the type of the product. The association between the number and type of the product will be collected by another operator on the basis of the association carried out by a dedicated software. The operator who will deliver the product will be informed about the type only at the end of the treatment.
  The data will be collected in pseudonymised form and inserted into a dedicated database in order to carry out the statistical analysis provided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hydrogen Peroxide and Hyaluronic acid (BMG0703) (Experimental): Patients will undergo a professional oral hygiene session (causal therapy) and will be instructed to perform proper oral hygiene manoeuvres at home.
  After the causal therapy, the treatment of the pockets will be performed by probing, between 3 and 7 mm, with BMG0703 by means of a dedicated sterile syringe. The application will be repeated after approx. 5 minutes.
  One bottle of BMG0703 will then be given to the patients who will be instructed to use it 3 times a day, after meals and after normal oral hygiene procedures, for at least one week.
  The subjects will then be re-evaluated after 3 days and after a week. During these check-ups, new samples will be collected at the level of the initial sampling sites and will be reassessed on the basis of the selected clinical indices (in particular plaque, bleeding and probing depth).
  Interventions: Drug: Hydrogen Peroxide and Hyaluronic acid filming formulation
- Chlorhexidine 0.2% (Active Comparator): Patients will undergo a professional oral hygiene session (causal therapy) and will be instructed to perform proper oral hygiene manoeuvres at home.
  After the causal therapy, the treatment of the pockets will be performed by probing, between 3 and 7 mm, with Chlorhexidine 0.2% by means of a dedicated sterile syringe. The application will be repeated after approx. 5 minutes.
  One bottle of Chlorhexidine 0.2% will then be given to the patients who will be instructed to use it 3 times a day, after meals and after normal oral hygiene procedures, for at least one week.
  The subjects will then be re-evaluated after 3 days and after a week. During these check-ups, new samples will be collected at the level of the initial sampling sites and will be reassessed on the basis of the selected clinical indices (in particular plaque, bleeding and probing depth).
  Interventions: Drug: Chlorhexidine 0.2%
- Placebo product (Placebo Comparator): Patients will undergo a professional oral hygiene session (causal therapy) and will be instructed to perform proper oral hygiene manoeuvres at home.
  After the causal therapy, the treatment of the pockets will be performed by probing, between 3 and 7 mm, with a placebo product by means of a dedicated sterile syringe. The application will be repeated after approx. 5 minutes.
  One bottle of the placebo product will then be given to the patients who will be instructed to use it 3 times a day, after meals and after normal oral hygiene procedures, for at least one week.
  The subjects will then be re-evaluated after 3 days and after a week. During these check-ups, new samples will be collected at the level of the initial sampling sites and will be reassessed on the basis of the selected clinical indices (in particular plaque, bleeding and probing depth).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydrogen Peroxide and Hyaluronic acid filming formulation — Patients will undergo a professional oral hygiene session (causal therapy) and will be instructed to perform proper oral hygiene manoeuvres at home.
  After the causal therapy, the treatment of the pockets will be performed by probing, between 3 and 7 mm, with BMG0703 by means of a dedicated sterile syringe. The application will be repeated after approx. 5 minutes.
  One bottle of BMG0703 will then be given to the patients who will be instructed to use it 3 times a day, after meals and after normal oral hygiene procedures, for at least one week.
  The subjects will then be re-evaluated after 3 days and after a week. During these check-ups, new samples will be collected at the level of the initial sampling sites and will be reassessed on the basis of the selected clinical indices (in particular plaque, bleeding and probing depth).
  Other Names: BMG0703
  Arms: Hydrogen Peroxide and Hyaluronic acid (BMG0703)
Drug: Chlorhexidine 0.2% — Patients will undergo a professional oral hygiene session (causal therapy) and will be instructed to perform proper oral hygiene manoeuvres at home.
  After the causal therapy, the treatment of the pockets will be performed by probing, between 3 and 7 mm, with Chlorhexidine 0.2% by means of a dedicated sterile syringe. The application will be repeated after approx. 5 minutes.
  One bottle of Chlorhexidine 0.2% will then be given to the patients who will be instructed to use it 3 times a day, after meals and after normal oral hygiene procedures, for at least one week.
  The subjects will then be re-evaluated after 3 days and after a week. During these check-ups, new samples will be collected at the level of the initial sampling sites and will be reassessed on the basis of the selected clinical indices (in particular plaque, bleeding and probing depth).
  Other Names: Chlorhexidine
  Arms: Chlorhexidine 0.2%
Drug: Placebo — Patients will undergo a professional oral hygiene session (causal therapy) and will be instructed to perform proper oral hygiene manoeuvres at home.
  After the causal therapy, the treatment of the pockets will be performed by probing, between 3 and 7 mm, with a placebo product by means of a dedicated sterile syringe. The application will be repeated after approx. 5 minutes.
  One bottle of the placebo product will then be given to the patients who will be instructed to use it 3 times a day, after meals and after normal oral hygiene procedures, for at least one week.
  The subjects will then be re-evaluated after 3 days and after a week. During these check-ups, new samples will be collected at the level of the initial sampling sites and will be reassessed on the basis of the selected clinical indices (in particular plaque, bleeding and probing depth).
  Other Names: Placebo product
  Arms: Placebo product

SUMMARY:
Assessment of the efficacy of BMG0703 in the treatment of periodontitis and control of supragingival plaque, compared to Chlorhexidine and a placebo product

DETAILED DESCRIPTION:
The enrolled subjects will be examined and treated by specialized medical personnel.

Patients will undergo a professional oral hygiene session (causal therapy) and will be instructed to perform proper oral hygiene manoeuvres at home.

Next, subjects will be divided into three groups: after the causal therapy, the treatment of the pockets will be performed by probing, between 3 and 7 mm, with the test product, active comparator or placebo, with the aid of a dedicated sterile syringe. The application will be repeated after approx. 5 minutes.

One bottle of the product (test, comparative or placebo) will then be given to the patient who will be instructed to use it 3 times a day, after meals and after normal oral hygiene procedures, for at least one week.

The subjects will then be re-evaluated after 3 days and after a week. During these check-ups, new samples will be collected at the level of the initial sampling sites and will be reassessed on the basis of the selected clinical indices (in particular plaque, bleeding and probing depth).

Patients with allergic reactions or hypersensitivity due to the use of the products will be advised to discontinue the use of the products and seek medical advice.

ELIGIBILITY:
Inclusion Criteria:

* Presence of periodontitis with pockets between 3 and 7 mm
* Acceptance of informed consent

Exclusion Criteria:

* subjects suffering from HIV
* subjects suffering from hepatitis
* serious systemic diseases preventing the use of specific dental therapies
* acute and/or chronic infectious pathologies
* inability to provide consent
* use of topical or systemic drugs
* inability to follow post-intervention hygiene instructions
* smokers

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Change in Bleeding index | 0, 3, 7, 30 days
  Subjects will undergo the measurement of bleeding index according to Silness J & Loe. Four surfaces per tooth (vestibular, lingual/palatal, mesial, distal) will be considered.
  Data will be collected based on four possible clinical conditions:
  Code 0: absence of bleeding during probing depth measurement; Code 1: absence of bleeding during probing depth measurement, presence of redness and oedema; Code 2: presence of bleeding during probing depth measurement with redness and oedema; Code 3: spontaneous bleeding
  Higher score means worse outcome.
Change in Plaque index | 0, 3, 7, 30 days
  Subjects will undergo the measurement of plaque index according to Silness J & Loe. Four surfaces per tooth (vestibular, lingual/palatal, mesial, distal) will be considered.
  Data will be collected based on four possible clinical conditions:
  Code 0: absence of plaque; Code 1: presence of plaque not visible to the naked eye but evidenced by the periodontal probe passage; Code 2: presence of plaque at the level of the gingival margin; Code 3: abundant presence of plaque at the level of the gingival margin and/or the rest of the dental surface.
  Higher score means worse outcome
  The sum of the values of the four surfaces examined, divided by the very number of surfaces, will give the plaque and bleeding index value for each individual tooth. The sum of the indices of each examined tooth divided by the total number of teeth examined will indicate the overall plaque and bleeding index of the subject at that time.

SECONDARY OUTCOMES:
Change in Microbiological analysis | 0,3,7,30 days
  The DNA-Sorb-B (Sacace) nucleic acid extraction kit will be used for the extraction and purification of bacterial DNA from clinical samples. Bacterial genome extraction is performed on 500 microlitres of oral sample fluid obtained from each patient.
  The molecular analysis, using Real Time PCR, involves the use of the KIT Periodontitis (PeriodontScreen Real-TM, Sacace), and in particular the following bacterial species will be researched: Porphyromonas gingivalis, Aggregatibacter actinomycetemcomitans, Treponema denticola, Fusobacterium nucleatum, Prevotella intermedia, Tannerella forsythia, Porphyromonas endodontalis.
  Periodontopathogenic bacteria are divided into high (Porphyromonas gingivalis, Aggregatibacter actinomycetemcomitans, Treponema denticle, Tannerella forsythia) and medium risk (Fusobacterium nucleatum, Prevotella Intermediate, Porphyromonas endodontalis). The results of the molecular analysis will be related to the clinical indices obtained from each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Giampietro Farronato, Professor, Principal Investigator — University of Milan; Gianguido Cossellu, Fellow, Principal Investigator — University of Milan
Locations (1):
- UOC Maxillofacial Surgery and Odontology, University of Milan, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data available upon request

REFERENCES:
- [Background] Caton J, Greenstein G, Polson AM. Depth of periodontal probe penetration related to clinical and histologic signs of gingival inflammation. J Periodontol. 1981 Oct;52(10):626-9. doi: 10.1902/jop.1981.52.10.626. PMID 6975365
- [Background] Fowler C, Garrett S, Crigger M, Egelberg J. Histologic probe position in treated and untreated human periodontal tissues. J Clin Periodontol. 1982 Sep;9(5):373-85. doi: 10.1111/j.1600-051x.1982.tb02048.x. PMID 6754765
- [Background] Polson AM, Caton JG, Yeaple RN, Zander HA. Histological determination of probe tip penetration into gingival sulcus of humans using an electronic pressure-sensitive probe. J Clin Periodontol. 1980 Dec;7(6):479-88. doi: 10.1111/j.1600-051x.1980.tb02154.x. PMID 6938528
- [Background] Keagle JG, Garnick JJ, Searle JR, King GE, Morse PK. Gingival resistance to probing forces. I. Determination of optimal probe diameter. J Periodontol. 1989 Apr;60(4):167-71. doi: 10.1902/jop.1989.60.4.167. PMID 2724029
- [Background] Hull PS, Clerehugh V, Ghassemi-Aval A. An assessment of the validity of a constant force electronic probe in measuring probing depths. J Periodontol. 1995 Oct;66(10):848-51. doi: 10.1902/jop.1995.66.10.848. PMID 8537866